CLINICAL TRIAL: NCT01964950
Title: Nesina Tablets Special Drug Use Surveillance Type 2 Diabetes Mellitus: Combination Therapy With Sulfonylurea
Brief Title: Alogliptin Tablets Special Drug Use Surveillance Type 2 Diabetes Mellitus: Combination Therapy With Sulfonylurea
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 121-013; JapicCTI-132266 (Registry Identifier: JapicCTI); JapicCTI-R160882 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-02

CONDITIONS: Surveillance
Keywords: drug therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alogliptin: All participants who received alogliptin 25 milligram (mg), tablets, orally, once daily for up to 12 months along with Sulfonylurea (SU) or without SU within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin as per routine clinical practice were observed in this study.

SUMMARY:
The purpose of this study is to examine the safety and efficacy of long-term combination therapy with alogliptin (Nesina) and sulfonylurea in participants with type 2 diabetes mellitus who responded inadequately to treatment with sulfonylurea in addition to diet therapy and exercise therapy.

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of alogliptin with a 1-year (12-month) observational period, designed to investigate the safety and efficacy of long-term combination therapy with alogliptin and sulfonylurea in participants with type 2 diabetes mellitus in a routine clinical setting.

Participants with type 2 diabetes mellitus who responded inadequately to treatment with sulfonylurea in addition to diet therapy and exercise therapy will be enrolled in this study. The planned sample size is 1,000.

The usual adult dosage for oral use is 1 alogliptin tablet (25 mg) once daily.

ELIGIBILITY:
Inclusion Criteria:

* Participants who did not adequately respond to the following treatment • Treatment with sulfonylurea in addition to diet therapy and exercise therapy

Exclusion Criteria:

1. Participants with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus (these participants require prompt adjustment of hyperglycemia by fluid infusion and insulin, and hence use of Nesina is not appropriate).
2. Participants with severe infection, pre- or post-operative participants, or participants with serious traumatic injury (blood glucose control by insulin injection is desirable for these participants, and hence use of Nesina is not appropriate).
3. Participants with a history of hypersensitivity to any ingredient of Nesina.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with type 2 diabetes mellitus who have been examined at a medical institution
Sampling Method: Non-Probability Sample
Enrollment: 1101 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda
Locations (1):
- Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 221 investigative sites in Japan from 1-Jul-11 to 31-Dec-14.
Pre-assignment Details: Participants with type 2 diabetes mellitus started treatment with alogliptin as per routine clinical practice were observed. As per protocol, participants we enrolled in 1 observational group at the start and were divided into 2 groups based on Sulfonylurea (SU) use for analysis of safety endpoints. Participant data was collected for overall arm.
Groups:
- All Population (Alogliptin): All participants who received alogliptin (Nesina) 25 milligram (mg), tablets, orally, once daily for up to 12 months along with an SU or without an SU within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin as per routine clinical practice were observed in this study.
Period: Overall Study
Arm/Group | All Population (Alogliptin)
Started | 1101 (Data reports overall population,since data not collected separately per arm as specified in protocol)
Completed | 1076
Not Completed | 25
Not completed — Protocol Violation | 25

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who completed the study and had safety data available.
Groups:
- Alogliptin + SU: Alogliptin (Nesina) 25 milligram (mg), tablets, orally, once daily for up to 12 months in participants who received an SU within 3 months from the start of administration of alogliptin and during the treatment period of alogliptin as per routine clinical practice were observed in this study.
- Alogliptin + Other: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months in participants who did not receive an SU within 3 months from the start of administration of alogliptin or during the treatment period of alogliptin as per routine clinical practice were observed in this study.
- Total: Total of all reporting groups
Arm/Group | Alogliptin + SU | Alogliptin + Other | Total
Number analyzed (Participants) | 916 | 160 | 1076
Age, Customized [Number; unit: participants]
  Less Than (<) 65 Years | 380 (11.67) | 69 (12.19) | 449
  Greater Than or Equal to (>=) 65 Years | 536 | 91 | 627
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 378 | 52 | 430
  Male | 538 | 108 | 646
Region of Enrollment [Number; unit: participants]
  Japan | 916 | 160 | 1076
Time From Diagnosis of Type 2 Diabetes [Number; unit: participants]
  Less than (<)2 years | 102 | 21 | 123
  Greater than or equal to (>=)2 to <5 years | 138 | 22 | 160
  >=5 to <10 years | 216 | 25 | 241
  >=10 years | 232 | 55 | 287
  Unknown | 228 | 37 | 265
Body Mass Index (BMI) [Number; unit: participants]
  <25 kilogram per square meter (kg/m^2) | 326 | 63 | 389
  >=25 kg/m^2 | 318 | 60 | 378
  Unknown | 272 | 37 | 309
Waist circumference [Number; unit: participants]
  <85 centimeter (cm) (Male) | 52 | 7 | 59
  >=85 cm (Male) | 102 | 22 | 124
  Unknown (Male) | 384 | 79 | 463
  <90 cm (Female) | 52 | 7 | 59
  >=90 cm (Female) | 39 | 4 | 43
  Unknown (Female) | 287 | 41 | 328
Pregnancy Status [Number; unit: participants] — This baseline characteristic was analyzed only in female participants.
  participants
    Not pregnant | 378 | 52 | 430
    Pregnant | 0 | 0 | 0
Healthcare Category [Number; unit: participants] — Participants were categorized as outpatient, inpatient, and outpatient and inpatient (participants who were both outpatient and inpatient during some point at the time and 3 months prior to enrollment).
  participants
    Outpatient | 891 | 156 | 1047
    Inpatient | 3 | 1 | 4
    Outpatient and Inpatient | 22 | 3 | 25
Degree of Renal Dysfunction [Number; unit: participants] — Estimated glomerular filtration rate (eGFR) was calculated using variables of gender, age at the start of treatment, and serum creatinine values, and severity was determined based on the following categories. If the serum creatinine value at the start of treatment was not listed, the severity was listed as "unknown." Normal: >=90 milliliter per minute (mL/min)/1.73^2, Mild: >=60 mL/min/1.73^2 to <90 mL/min/1.73^2 Moderate: >=30 mL/min/1.73^2 to <60 mL/min/1.73^2, Severe: <30 mL/min/1.73^2. eGFR = 194 * Cr^-1.094 * (age)^-0.287 (* 0.739 if female), where Cr is serum creatinine
  participants
    Normal | 151 | 25 | 176
    Mild | 351 | 61 | 412
    Moderate | 146 | 25 | 171
    Severe | 12 | 0 | 12
    Unknown | 256 | 49 | 305
History of Allergy [Number; unit: participants]
  Did not have allergy | 742 | 131 | 873
  Had allergy | 78 | 8 | 86
  Unknown | 96 | 21 | 117
Health-related Complications [Number; unit: participants]
  Had complications | 837 | 145 | 982
  Had no complications | 79 | 15 | 94
Diabetic Complications [Number; unit: participants]
  Had complications | 187 | 43 | 230
  Had no complications | 729 | 117 | 846
Breakdown of Diabetic Complications [Number; unit: participants] — This baseline characteristic was analyzed only in participants who had diabetic complications. Participants may be represented in more than 1 category.
  participants
    Diabetic nephropathy | 114 | 23 | 137
    Diabetic retinopathy | 76 | 21 | 97
    Diabetic neuropathy | 61 | 20 | 81
Complications of Hypertension [Number; unit: participants]
  Had complications | 593 | 97 | 690
  Had no complications | 323 | 63 | 386
Complications of Dyslipidemia [Number; unit: participants]
  Had complications | 582 | 99 | 681
  Had no complications | 334 | 61 | 395
Complications of Hyperuricemia [Number; unit: participants]
  Had complications | 74 | 8 | 82
  Had no complications | 842 | 152 | 994
Complications of Liver Damage [Number; unit: participants]
  Had complications | 181 | 35 | 216
  Had no complications | 735 | 125 | 860
Breakdown of Complications of Liver Damage [Number; unit: participants] — Liver damage complications were categorized as hepatic steatosis, hepatitis alcoholic, chronic hepatitis, hepatic cirrhosis and any other complications related to liver damage. This baseline characteristic was analyzed only in participants who had complications of liver damage. Participants may be represented in more than 1 category.
  participants
    Hepatic steatosis | 122 | 24 | 146
    Hepatitis alcoholic | 30 | 9 | 39
    Chronic hepatitis | 31 | 5 | 36
    Hepatic cirrhosis | 2 | 1 | 3
    Other | 4 | 0 | 4
Degree of Hepatic Dysfunction [Number; unit: participants] — Severity was determined using aspartate aminotransferase (AST) or alanine transaminase (ALT) values at the start of treatment with alogliptin. For the assessment of severity, the following categories were used and a higher severity grade for either AST or ALT serum levels was adopted. Normal: <50 international units per liter (IU/L), Grade 1: >=50 to <100 IU/L, Grade 2: >=100 to <500 IU/L, and Grade 3: >=500 IU/L.
  participants
    Normal | 599 | 111 | 710
    Grade 1 | 75 | 11 | 86
    Grade 2 | 10 | 2 | 12
    Unknown | 232 | 36 | 268
Complications of Renal Damage [Number; unit: participants]
  Had complications | 126 | 27 | 153
  Had no complications | 790 | 133 | 923
Breakdown of Complications of Renal Damage [Number; unit: participants] — Renal damage complications were categorized as nephrotic syndrome, glomerulonephritis, renal failure chronic and any other complications related to renal damage. This baseline characteristic was analyzed only in participants who had renal damage complications. Participants may be represented in more than 1 category.
  participants
    Nephrotic syndrome | 3 | 1 | 4
    Glomerulonephritis | 2 | 1 | 3
    Renal failure chronic | 9 | 0 | 9
    Other | 113 | 25 | 138
Complications of Heart Disease [Number; unit: participants]
  Had complications | 129 | 18 | 147
  Had no complications | 787 | 142 | 929
Breakdown of Complications of Heart Disease [Number; unit: participants] — Heart disease complications were categorized as cardiac failure, myocardial infarction, angina pectoris, and any other complications related to heart disease. This baseline characteristic was analyzed only in participants who had heart disease complications. Participants may be represented in more than 1 category.
  participants
    Cardiac failure | 25 | 3 | 28
    Myocardial infarction | 26 | 4 | 30
    Angina pectoris | 70 | 7 | 77
    Other | 26 | 4 | 30
Complications of Heart Failure [Number; unit: participants]
  Had complications | 25 | 3 | 28
  Had no complications | 891 | 157 | 1048
New York Heart Association (NYHA) Heart Failure Classification [Number; unit: participants] — NYHA functional classification ranges from Class I (participants with cardiac disease but without resulting limitations of physical activity), Class II (participants with cardiac disease resulting in slight limitation of physical activity), Class III (participants with cardiac disease resulting in marked limitation of physical activity), Class IV (participants with cardiac disease resulting in inability to carry on any physical activity without discomfort). This baseline measure was analyzed only for participants who had complications of heart failure.
  participants
    NYHA Class I | 16 | 2 | 18
    NYHA Class II | 5 | 0 | 5
    NYHA Class III | 1 | 0 | 1
    NYHA Class IV | 1 | 0 | 1
    Unknown | 2 | 1 | 3
Complications of Stroke-related Disease [Number; unit: participants]
  Had complications | 65 | 7 | 72
  Had no complications | 851 | 153 | 1004
Breakdown of Complications of Stroke-related Disease [Number; unit: participants] — This baseline characteristic was analyzed only in participants who had complications of stroke-related disease.
  participants
    Cerebral infarction | 64 | 7 | 71
    Cerebral haemorrhage | 1 | 0 | 1
Complications of Allergic Disease [Number; unit: participants]
  Had complications | 51 | 7 | 58
  Had no complications | 865 | 153 | 1018
Complications of Malignant Tumor [Number; unit: participants]
  Had complications | 19 | 3 | 22
  Had no complications | 897 | 157 | 1054
Presence of Medical History [Number; unit: participants]
  Had medical history | 165 | 31 | 196
  Did not have medical history | 652 | 113 | 765
  Unknown | 99 | 16 | 115
History of Alcohol Consumption [Number; unit: participants] — In this measure, participants responded whether they consumed alcohol-containing beverages nearly every day or not.
  participants
    Yes | 228 | 44 | 272
    No | 527 | 84 | 611
    Unknown | 161 | 32 | 193
Smoking Classification [Number; unit: participants]
  Never smoked | 372 | 51 | 423
  Current smoker | 145 | 30 | 175
  Ex-smoker | 189 | 39 | 228
  Unknown | 210 | 40 | 250
Glycosylated Hemoglobin (HbA1c) Level [Number; unit: participants]
  HbA1c <6.0 percent (%) | 14 | 4 | 18
  HbA1c >=6.0% to <7.0% | 149 | 25 | 174
  HbA1c >=7.0% to <8.0% | 312 | 61 | 373
  HbA1c >=8.0% | 374 | 61 | 435
  Unknown | 67 | 9 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. The safety analysis was planned to be assessed in alogliptin + SU and alogliptin + other arm separately.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who completed the study and had safety data available.
Measure: Number; unit: participants
Arm/Group | Alogliptin + SU | Alogliptin + Other
Number analyzed (Participants) | 916 | 160
participants | 19 | 1

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reaction
Description: Serious adverse drug reactions are defined as serious adverse events (SAEs) which are in the investigator's opinion of causal relationship to the study treatment. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The safety analysis was planned to be assessed in alogliptin + SU and alogliptin + other arm separately.
Time Frame: Baseline up to 12 months
Population: The safety analysis set was defined as all participants who completed the study and had safety data available.
Measure: Number; unit: participants
Arm/Group | Alogliptin + SU | Alogliptin + Other
Number analyzed (Participants) | 916 | 160
participants | 5 | 0

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of SU treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Groups:
- Alogliptin: Participants who took alogliptin 25 mg, tablets, orally, once daily for up to 12 months as per routine clinical practice were observed.
Arm/Group | Alogliptin
Number analyzed (Participants) | 830
percentage of glycosylated hemoglobin
  Baseline (n=830) | 8.03 (1.348)
  Change at Month 1 (n = 655) | -0.40 (0.708)
  Change at Month 3 (n = 710) | -0.66 (1.117)
  Change at Month 6 (n = 725) | -0.72 (1.117)
  Change at Month 12 (n = 670) | -0.64 (1.106)
  Change at Final Assessment (n = 830) | -0.65 (1.145)

4. Secondary Outcome: Percentage of Participants Achieving Objective Glycemic Control
Description: The rate of achieving objective glycemic control in HbA1c level was calculated at baseline and final visit (last visit for a participant in the study, up to Month 12). Glycemic control was measured as <8.0%, <7.0%, and <6.0% of glycosylated hemoglobin. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of SU treatment.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin
Number analyzed (Participants) | 830
percentage of participants
  <8.0 percent: Baseline | 56.3
  <8.0%: Final Assessment | 75.4
  <7.0%: Baseline | 19.3
  <7.0%: Final Assessment | 43.0
  <6.0%: Baseline | 1.7
  <6.0%: Final Assessment | 4.6

5. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The change between the fasting blood glucose value collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of the SU treatment.
Time Frame: Baseline, Months 1, 3, 6, 12, and final assessment (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had fasting blood glucose data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Alogliptin
Number analyzed (Participants) | 250
milligram per deciliter (mg/dL)
  Baseline (n = 250) | 151.1 (43.07)
  Change at Month 1 (n = 159) | -14.6 (42.91)
  Change at Month 3 (n = 175) | -13.8 (40.08)
  Change at Month 6 (n = 185) | -13.1 (47.37)
  Change at Month 12 (n = 168) | -16.4 (43.97)
  Change at Final Assessment (n = 250) | -13.7 (49.10)

6. Secondary Outcome: Change From Baseline in Fasting Insulin Level
Description: The change between the fasting insulin value collected at 1 month, 3 months, 6 months, 12 months or final visit (last visit for a participant in the study, up to Month 12) relative to baseline. The efficacy analysis was planned to be assessed in the total alogliptin arm irrespective of SU treatment.
Time Frame: Months 1, 3, 6, 12, and final assessment (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had fasting insulin data at baseline and post-baseline time points available.
Measure: Mean (Standard Deviation); unit: micro units per milliliter (mcU/mL)
Arm/Group | Alogliptin
Number analyzed (Participants) | 33
micro units per milliliter (mcU/mL)
  Baseline (n = 33) | 7.88 (5.674)
  Change at Month 1 (n = 15) | 1.27 (12.138)
  Change at Month 3 (n = 17) | 0.21 (3.474)
  Change at Month 6 (n = 20) | 0.69 (5.629)
  Change at Month 12 (n = 22) | 1.17 (3.521)
  Change at Final Assessment (n = 33) | 1.86 (5.455)

ADVERSE EVENTS:
Time Frame: Baseline up to 12 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were collected in the safety population.
Arm/Group | Alogliptin + SU | Alogliptin + Other
Serious Adverse Events (participants affected / at risk) | 5/916 | 0/160
Other Adverse Events (participants affected / at risk) | 19/916 | 1/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin + SU (N=916) | Alogliptin + Other (N=160)
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin + SU (N=916) | Alogliptin + Other (N=160)
Influenza (Infections and infestations) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Feeling abnormal (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.